CLINICAL TRIAL: NCT01346761
Title: Bridging Geographic Barriers: Remote Cancer Genetic Counseling for Rural Women
Brief Title: Risk Education and Assessment for Cancer Heredity
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anita Kinney, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23146; 1R01CA129142-01A2 (NIH)
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer; Ovarian Cancer; Genetic Predisposition
Keywords: Genetic Counseling; Genetic Counseling Interventions; Genetic Testing; BRCA1 gene; BRCA2 gene; Risk Communication
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Genetic Predisposition to Disease; Fanconi Anemia, Complementation Group D1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone genetic counseling (Experimental): Participants randomly assigned to telephone counseling are mailed packets that included a sealed envelope containing an educational brochure about hereditary breast and ovarian cancer (HBOC) genetic counseling with visual aids. At the time of their session, participants open their envelope and counselors use the visual aids to explain breast-ovarian cancer genetics and administer BRCA1/BRCA2 genetic counseling. Women receiving in-person counseling are given these same materials during their session at the community clinic. In-person and telephone counseling are delivered by the same five board-certified genetic counselors.
  Interventions: Behavioral: Telephone Genetic Counseling
- In-person genetic counseling (Active Comparator): In-person BRCA1/BRCA2 genetic counseling is delivered by board-certified genetic counselors using a guide-line-concordant semistructured protocol that allows for personalization of counseling and is similar to that used by others. All sessions are audiotaped for treatment fidelity assessments. In-person and telephone counseling are delivered by the same five board-certified genetic counselors.
  Interventions: Behavioral: In-Person Genetic Counseling

INTERVENTIONS:
Behavioral: Telephone Genetic Counseling — Participants will complete a pre-test session and a test results disclosure session (if tested) with a licensed, board-certified genetic counselor over the telephone. Counseling sessions will be audiotaped for quality control of intervention.
  Other Names: BRCA1/BRCA2 genetic counseling via telephone
  Arms: Telephone genetic counseling
Behavioral: In-Person Genetic Counseling — Participants will complete a pre-test session and a test results disclosure session (if tested) with a licensed, board-certified genetic counselor in person. Counseling sessions will be audiotaped for quality control of intervention.
  Other Names: BRCA1/BRCA2 traditional genetic counseling in-person
  Arms: In-person genetic counseling

SUMMARY:
Individuals living in geographically underserved areas encounter considerable barriers to access of quality cancer genetic services. Although in-person genetic counseling has generally been accepted as the standard of care, the use of telecommunications to deliver clinical genetic services may help reduce this disparity in access to such services. However, before the widespread adoption of telephone-delivered cancer genetic services occurs, it is critical to analyze the efficacy and safety of this mode of communication. This two-group randomized equivalency/non-inferiority trial will determine whether telephone-based cancer genetic counseling is an acceptable alternative to the traditional in-person mode among women who have a personal or family history of breast and/or ovarian cancer strong enough to warrant genetic counseling and testing. This study's findings will provide important information to cancer centers and cancer control policies about the safety, efficacy, and costs of delivering telephone-based clinical cancer genetic services for geographically challenged women at risk for having Breast Cancer susceptibility gene (BRCA) 1/2 mutations.

DETAILED DESCRIPTION:
Following confirmation of eligibility and completion of baseline surveys, participants will be randomly assigned to one of the study arms by the project coordinator, using a computer-generated allocation algorithm on the basis of a randomization blocks method using four, six or eight participants in each block.

In-person and telephone counseling will be delivered by the same board-certified genetic counselors using a guideline-concordant semi-structured protocol that will allow for personalization of counseling.

Participants randomly assigned to telephone counseling will be mailed packets that include a sealed envelope containing an educational brochure about hereditary breast and ovarian cancer genetic counseling with visual aids. At the time of their session, participants will review the brochure and genetic counselors will use visual aids to explain breast-ovarian cancer genetics. Women receiving in-person counseling will be given the same materials during their session at the community clinic.

For women who elect to have testing, those who have telephone counseling will be sent a genetic test kit; those who have in-person counseling will have the option of giving a sample immediately at the clinic, or will be given a test kit with the same instructions as those in the telephone-counseling group.

When BRCA test results become available, participants will be offered individual post-test counseling with the same genetic counselor who conducted the pretest session.

ELIGIBILITY:
Inclusion Criteria:

* Utah resident
* Meets National Comprehensive Cancer Network (NCCN) guidelines for hereditary breast/ovarian cancer syndrome (personal and/or family history of breast and/or ovarian cancer, or is a member of a family with a known positive BRCA1/BRCA2 mutation).

Exclusion Criteria:

* Has had genetic counseling and/or BRCA 1/2 testing
* Physically or mentally unable to complete telephone surveys, telephone or in-person counseling or provide informed consent.
* Unable to read and speak English fluently
* Unable to travel to in-person genetic counseling session (17 in-person sites throughout Utah)
* Male gender

Ages: 25 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determine the non-inferiority/equivalency of telephone genetic counseling to standard in-person genetic counseling | 6 &12-month follow-up
  1. Compare utilization of BRCA1/BRCA2 testing among telephone genetic counseling relative to in-person genetic counseling.
  2. Determine the safety and efficacy of telephone genetic counseling relative to in-person genetic counseling by evaluating psychological and quality of life outcomes.
  3. Compare communication-related and decision-making outcomes among telephone genetic counseling relative to in-person genetic counseling.

SECONDARY OUTCOMES:
Determine the feasibility of the intervention | 1 week pre-test, 1 week post-test, 6 & 12 month follow-ups
  1. Examine the intervention delivery and patient costs of telephone genetic counseling relative to in-person genetic counseling.
  2. Examine mediators (sociodemographic, communication factors, health care access, clinical, & psychosocial factors) of genetic testing decisions, and affective and cognitive outcomes.
  3. Compare decisions and perceptions about use of primary/secondary prevention strategies for hereditary breast/ovarian cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y. Kinney, R.N., Ph.D., Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Steffen LE, Du R, Gammon A, Mandelblatt JS, Kohlmann WK, Lee JH, Buys SS, Stroup AM, Campo RA, Flores KG, Vicuna B, Schwartz MD, Kinney AY. Genetic Testing in a Population-Based Sample of Breast and Ovarian Cancer Survivors from the REACH Randomized Trial: Cost Barriers and Moderators of Counseling Mode. Cancer Epidemiol Biomarkers Prev. 2017 Dec;26(12):1772-1780. doi: 10.1158/1055-9965.EPI-17-0389. Epub 2017 Sep 29. PMID 28971986
- [Derived] Kinney AY, Steffen LE, Brumbach BH, Kohlmann W, Du R, Lee JH, Gammon A, Butler K, Buys SS, Stroup AM, Campo RA, Flores KG, Mandelblatt JS, Schwartz MD. Randomized Noninferiority Trial of Telephone Delivery of BRCA1/2 Genetic Counseling Compared With In-Person Counseling: 1-Year Follow-Up. J Clin Oncol. 2016 Aug 20;34(24):2914-24. doi: 10.1200/JCO.2015.65.9557. Epub 2016 Jun 20. PMID 27325848